CLINICAL TRIAL: NCT06984692
Title: Evaluation of iRise mHealth App on Healthcare Workers' (HCWs') Self-Efficacy and Willingness to Respond During Public Health Emergencies in Pakistan
Acronym: iRise
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to collaboration model change
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00029867; 5R33TW012210-04 (NIH)
Record Dates: First submitted 2025-05-08; First posted 2025-05-22 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Behavior Change; Self Efficacy

STUDY DESIGN:
Intervention Model Description: This will be a 12-month, two-arm, parallel randomized controlled trial to evaluate a mHealth intervention, iRise, for emergency health care workers (HCWs).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Curriculum (Active Comparator): Control group: The control group will receive standard training in crisis response and management, which is offered as a course on Emergency Management and Response at AKU, for which study participants from JPMC will also readily access. Participants will be able to both view and download the course content via internet and can request a printed version of the course. The course involves introduction to disaster terminology, emergency management cycle and hospital-based patient treatment guidelines. The control curriculum will offer a comprehensive focus on disaster preparedness, addressing important subjects such as emergency management techniques, disasters, and triage. The eight-hour training will be split into two parts, aiming to improve academic and practical understanding. The first part will be a didactic session, where participants will learn fundamental information through lectures and discussions. The second part will consist of hands-on training.
  Interventions: Other: Control Curriculum
- iRise curriculum (Experimental): The intervention group would download the iRise mHealth app ("iRise app") via Canvas on the participant's respective smart phones, and based on the participant's own schedules and preferences, would complete different modules of iRise. The iRise app would include emergency management elements as received by the control group, but presented via smart phone-based content delivery (i.e., rather than rather than via the in-person modality utilized for the control group).
  Interventions: Other: iRise curriculum

INTERVENTIONS:
Other: iRise curriculum — Intervention group: The intervention group would download the iRise mHealth app ("iRise app") via Canvas on the participant's respective smart phones, and based on the participant's own schedules and preferences, would complete different modules of iRise. The iRise app would include emergency management elements as received by the control group, but presented via smart phone-based content delivery (i.e., rather than rather than via the in-person modality utilized for the control group).
  Arms: iRise curriculum
Other: Control Curriculum — The control group will receive standard training in crisis response and management, which is offered as a course on Emergency Management and Response at AKU, for which study participants from JPMC will also readily access. The course involves introduction to disaster terminology, emergency management cycle and hospital-based patient treatment guidelines. The control curriculum will offer a comprehensive focus on disaster preparedness, addressing important subjects such as emergency management techniques, disasters, and triage. The eight-hour training will be split into two parts, aiming to improve academic and practical understanding. The first part will be a didactic session, where participants will learn fundamental information through lectures and discussions. The second part will consist of hands-on training, allowing attendees to practice and apply learned concepts in simulated emergency scenarios.
  Arms: Control Curriculum

SUMMARY:
The purpose of this study is to assess the effectiveness of a novel mHealth intervention that is being designed to promote self-efficacy and response willingness among Pakistan-based emergency department health care workers (HCWs) in public health emergencies and disasters. This application seeks approval for the trial of the intervention. The purpose of this trial is to gauge short-term (1-month), medium-term (6-months), and longer-term (12-months) impacts of iRise mHealth app on low and middle income based countries HCWs' self-efficacy and willingness to respond (WTR) during public health emergencies and disasters. The investigators will test the hypothesis that the iRise app would yield an increased 12-months WTR in Aga Khan University Hospital (AKUH) and Jinnah Postgraduate Medical Center (JMPC) emergency departments.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study if

* aged 18 years or older,
* have worked in the current job position for at least three months,
* current Emergency Department clinical staff/employee involved in direct patient care (doctors, nurses, and technicians) at a participating institution (Aga Khan University Hospital (AKUH), Jinnah Postgraduate Medical Centre (JPMC)
* understand and write English,
* own a smart phone and have access to the internet to download the app.

Exclusion Criteria:

Participants will not be eligible to participate if

* younger than 18 years of age,
* have worked in the current job position for less than three months,
* are not a current employee or staff member as described above,
* are auxiliary personnel such as registration staff, housekeeping, porters, and security personnel,
* don't understand and write English, or
* don't own a smart phone or have access to the internet to download the app.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Willingness to respond (WTR) to disasters as measured by Hospital Infrastructure Response Survey Tool (HIRST) | Baseline, 1 month, 6 months, 12 months
  HIRST uses a 9-point Likert scale [1= Strongly Agree; 9 = Strongly Disagree] or "Don't Know) to indicate attitudes and beliefs about a series of 20 construct statements relevant to emergency response risk perception. Score range 20-180. Higher scores indicate a greater willingness to respond or preparedness.
Willingness to respond (WTR) to disasters as measured by Hospital Infrastructure Response Survey Tool (HIRST) | 1 month
  HIRST uses a 9-point Likert scale [1= Strongly Agree; 9 = Strongly Disagree] or "Don't Know) to indicate attitudes and beliefs about a series of 20 construct statements relevant to emergency response risk perception. Score range 20-180. Higher scores indicate a greater willingness to respond or preparedness.
Willingness to respond (WTR) to disasters as measured by Hospital Infrastructure Response Survey Tool (HIRST) | 6 months
  HIRST uses a 9-point Likert scale [1= Strongly Agree; 9 = Strongly Disagree] or "Don't Know) to indicate attitudes and beliefs about a series of 20 construct statements relevant to emergency response risk perception. Score range 20-180. Higher scores indicate a greater willingness to respond or preparedness.
Willingness to respond (WTR) to disasters as measured by Hospital Infrastructure Response Survey Tool (HIRST) | 12 months
  HIRST uses a 9-point Likert scale [1= Strongly Agree; 9 = Strongly Disagree] or "Don't Know) to indicate attitudes and beliefs about a series of 20 construct statements relevant to emergency response risk perception. Score range 20-180. Higher scores indicate a greater willingness to respond or preparedness.

SECONDARY OUTCOMES:
Self efficacy as assessed by the General Self-efficacy Scale | Baseline
  Self efficacy is assessed by the General Self-efficacy Scale embedded within the Hospital Infrastructure Response Survey Tool (HIRST).Total score ranging between 10 and 40, with a higher score indicating a higher level of self efficacy
Self efficacy as assessed by the General Self-efficacy Scale | 1 month
  Self efficacy is assessed by the General Self-efficacy Scale embedded within the Hospital Infrastructure Response Survey Tool (HIRST).Total score ranging between 10 and 40, with a higher score indicating a higher level of self efficacy
Self efficacy as assessed by the General Self-efficacy Scale | 6 months
  Self efficacy is assessed by the General Self-efficacy Scale embedded within the Hospital Infrastructure Response Survey Tool (HIRST).Total score ranging between 10 and 40, with a higher score indicating a higher level of self efficacy
Self efficacy as assessed by the General Self-efficacy Scale | 12 months
  Self efficacy is assessed by the General Self-efficacy Scale embedded within the Hospital Infrastructure Response Survey Tool (HIRST).Total score ranging between 10 and 40, with a higher score indicating a higher level of self efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Barnett, MD, Principal Investigator — Johns Hopkins University
Locations (3):
- Pakistan (3):
  - Aga Khan University Hospital, Karachi, Sindh
  - Jinnah Postgraduate Medical Centre, Karachi, Sindh
  - Aga khan university, Karachi, Sindh

IPD SHARING:
Plan to Share IPD: No